CLINICAL TRIAL: NCT04645823
Title: Spinal Fentanyl or Epidural Analgesia in the Early First Phase of Induced Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Women's Hospital HUS (Other)
Responsible Party: Principal Investigator, Antti Vaananen, Anesthesiologist, Women's Hospital HUS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Versio4_22112020; 2020-005506-26 (EudraCT Number)
Record Dates: First submitted 2020-11-22; First posted 2020-11-27 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Labor Pain; Induced; Birth
Keywords: epidural analgesia; spinal analgesia; labor pain
MeSH Terms: conditions — Labor Pain | interventions — Fentanyl; Lidocaine

STUDY DESIGN:
Intervention Model Description: 60 parturients randomized to two different treatment arms (30 in each group)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The parturient and the midwife as well as the researcher doing the interview for analgesia will be masked. The anesthesiologist performing either spinal fentanyl administration or epidural analgesia will not be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spinal fentanyl (Active Comparator): Using a combined spinal epidural technique a single dose of 20 µg of fentanyl diluted into 2 ml with NaCl 0.9 % will be injected into the CSF at lower lumbar interspace. An epidural catheter is left in place for subsequent analgesic doses.
  Interventions: Drug: Fentanyl Citrate
- Epidural lidocaine and fentanyl (Experimental): Using a catheter in the epidural space in the lower lumbar interspace a single dose of lidocaine (80 mg) and fentanyl (100 µg) is given. The epidural catheter is left in place for subsequent analgesic doses.
  Interventions: Drug: Lidocaine 1% Injectable Solution; Drug: Fentanyl Citrate

INTERVENTIONS:
Drug: Fentanyl Citrate — Fentanyl citrate 20 µg in 2 ml of saline injected into csf
  Arms: Spinal fentanyl
Drug: Lidocaine 1% Injectable Solution — Fentanyl citrate 100µg and lidocaine hydrochloride 80 mg in 10 ml volume
  Arms: Epidural lidocaine and fentanyl
Drug: Fentanyl Citrate — Fentanyl citrate 100µg and lidocaine hydrochloride 80 mg in 10 ml volume
  Arms: Epidural lidocaine and fentanyl

SUMMARY:
A total of 60 parturients undergoing induction of labour will be consented to participate in the study where they will be randomized to receive either spinal fentanyl (20 µg) or epidural analgesia (fentanyl 100µg and lidocaine 80 mg).

They will be monitored for the development of analgesia for a duration of 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Signs a consent form to participate voluntarily into the trial
2. Induced labor
3. singleton pregnancy
4. primiparous
5. BMI 20-40 at the time of delivery
6. No history of allergy for lidocaine or fentanyl
7. sufficient command of Finnish language to understand the consent form and interview
8. Cervical dilatation at maximum 4 cm at the time of intervention

Exclusion Criteria:

1. Any contraindication for spinal or epidural analgesia
2. Allergy for lidocaine or fentanyl
3. The patient has received any opioid medication within 90 minutes prior to intervention

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All recruited patients are parturients undergoing induction of labor
Enrollment: 60 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Analgesia at 20 minutes | 20 minutes
  Reduction of visual analog scale (VAS) pain during contraction from pre-intervention value. 0 mm means no pain while 100 mm means worst possible pain.

SECONDARY OUTCOMES:
Time until pain returns to 60 mm VAS | 30-180 minutes
  Time from intervention until the maximum pain during contraction return to 60 mm on VAS scale
Ambulation during the analgesia provided by the intervention | 30-180 minutes
  HAs the parturient been walking during the analgesia provided by the intervention
Changes in the cardiotocography (fetal heart rate) within 30 minutes after the intervention | 0-30 minutes
  Graded as normal, susceptible, pathological
Pruritus | 0-30 minutes
  The incidence of pruritus within 30 minutes after the intervention, graded: none, mild, moderate, severe, unbearable
SAtisfaction of the parturient with the analgesia provided by the intervention | at 30 minutes
  On 0-100 mm visual analog scale (VAS). Where 0 means no satisfaction at all and 100 mm means maximum satisfaction.
Cervical dilatation rate cm/h during the analgesia intervention | 0-180 min
  (The cervical dilatation (1-10 cm) 1-3 hours post analgesia - The cervical dilatation (1-5 cm) before analgesia) / time between measurements (hours)
Use of oxytocin during the analgesia study period | 30 min
  Oxytocin administered i.v. during 0-30 minutes after the analgesia (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Antti J Vaananen, MD PhD, Principal Investigator — HUCH, Women's hospital/dept of anesthesia
Locations (1):
- HUS/Women's hospital dept of anaesthesia, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salmi L, Jernman R, Vaananen A. Is epidural analgesia non-inferior to intrathecal fentanyl as initiation for neuraxial analgesia in early non-spontaneous labour? Acta Anaesthesiol Scand. 2024 May;68(5):664-674. doi: 10.1111/aas.14389. Epub 2024 Feb 16. PMID 38366324